CLINICAL TRIAL: NCT00871949
Title: A Phase 1 Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of PNU-100480 (PF-02341272) After First Time Administration Of Ascending Oral Doses To Healthy Adult Subjects Under Fed And Fasted Conditions
Brief Title: Safety, Tolerability And Pharmacokinetics Study Of Single Doses Of PNU-100480 In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sequella, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B1171001
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Tuberculosis
Keywords: Safety tolerability pharmacokinetics PK first in human FIH
MeSH Terms: conditions — Tuberculosis | interventions — PNU-100480

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1, Sequence 1 (Experimental): Period 1- Placebo Period 2- 100 mg Period 3- 300 mg
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 1, Sequence 2 (Experimental): Period 1- 35 mg Period 2- Placebo Period 3- 300 mg
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 1, Sequence 3 (Experimental): Period 1- 35 mg Period 2- 100 mg Period 3- Placebo
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 2, Sequence 1 (Experimental): Period 1- Placebo Period 2- 1000 mg Period 3- 1500 mg Period 4- 600 mg (Fed conditions)
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 2, Sequence 2 (Experimental): Period 1- 600 mg Period 2- Placebo Period 3- 1500 mg Period 4- 600 mg (Fed conditions)
  Interventions: Drug: PNU-100480; Drug: Placebo
- Cohort 2, Sequence 3 (Experimental): Period 1- 600 mg Period 2- 1000 mg Period 3- Placebo Period 4- 600 mg (Fed conditions)
  Interventions: Drug: PNU-100480; Drug: Placebo

INTERVENTIONS:
Drug: PNU-100480 — 100 mg oral suspension given once
  Other Names: Period 2
  Arms: Cohort 1, Sequence 1
Drug: PNU-100480 — 300 mg oral suspension given once
  Other Names: Period 3
  Arms: Cohort 1, Sequence 1
Drug: Placebo — placebo to match oral suspension given once
  Other Names: Period 1
  Arms: Cohort 1, Sequence 1
Drug: PNU-100480 — 300 mg oral suspension given once
  Other Names: Period 3
  Arms: Cohort 1, Sequence 2
Drug: PNU-100480 — 35 mg oral suspension given once
  Other Names: Period 1
  Arms: Cohort 1, Sequence 2
Drug: Placebo — placebo to match oral suspension given once
  Other Names: Period 2
  Arms: Cohort 1, Sequence 2
Drug: PNU-100480 — 100 mg oral suspension given once
  Other Names: Period 2
  Arms: Cohort 1, Sequence 3
Drug: PNU-100480 — 35 mg oral suspension given once
  Other Names: Period 1
  Arms: Cohort 1, Sequence 3
Drug: Placebo — placebo to match oral suspension given once
  Other Names: Period 3
  Arms: Cohort 1, Sequence 3
Drug: PNU-100480 — 1000 mg oral suspension given once
  Other Names: Period 2
  Arms: Cohort 2, Sequence 1
Drug: PNU-100480 — 1500 mg oral suspension given once
  Other Names: Period 3
  Arms: Cohort 2, Sequence 1
Drug: PNU-100480 — Fed conditions, 600 mg oral suspension given once
  Other Names: Period 4 (Fed)
  Arms: Cohort 2, Sequence 1
Drug: Placebo — placebo to match oral suspension given once
  Other Names: Period 1
  Arms: Cohort 2, Sequence 1
Drug: PNU-100480 — 1500 mg oral suspension given once
  Other Names: Period 3
  Arms: Cohort 2, Sequence 2
Drug: PNU-100480 — 600 mg oral suspension given once
  Other Names: Period 1
  Arms: Cohort 2, Sequence 2
Drug: PNU-100480 — Fed conditions, 600 mg oral suspension given once
  Other Names: Period 4 (Fed)
  Arms: Cohort 2, Sequence 2
Drug: Placebo — placebo to match oral suspension given once
  Other Names: Period 2
  Arms: Cohort 2, Sequence 2
Drug: PNU-100480 — 1000 mg oral suspension given once
  Other Names: Period 2
  Arms: Cohort 2, Sequence 3
Drug: PNU-100480 — 600 mg oral suspension given once
  Other Names: Period 1
  Arms: Cohort 2, Sequence 3
Drug: PNU-100480 — Fed conditions, 600 mg oral suspension given once
  Other Names: Period 4 (Fed)
  Arms: Cohort 2, Sequence 3
Drug: Placebo — placebo to match oral suspension given once
  Other Names: Period 3
  Arms: Cohort 2, Sequence 3

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of PNU-100480 (PF-02341272) after a single dose in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers willing and able to be confined to the Clinical Research Unit and comply with study schedule.
* Women of non-childbearing potential only.

Exclusion Criteria:

* History of hypersensitivity to, or intolerance of, linezolid.
* Antibiotic treatment within 14 days prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability of escalating single oral doses of PNU-100480. | Daily, Days 1-3 or 4, and 7-14 days after dosing.

SECONDARY OUTCOMES:
Characterize pharmacokinetics of single oral doses PNU-100480. | Predose; multiple timepoints postdose on Day 1, and up to 72 hours postdose.
Characterize the effect of food on the pharmacokinetics of a single oral dose of PNU-100480. | Predose; multiple timepoints postdose on Day 1, and up to 72 hours postdose.
Characterize the bactericidal activity in blood of orally administered PNU-100480 against intracellular Mycobacterium tuberculosis in relation to blood concentrations of PNU-100480 (and its metabolites) (some periods only) | Predose and timpoints up to 24 hours post dose on Day 1 (only in some periods)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Beth Ferstenberg, M.D., Study Director — Sequella, Inc.
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Wallis RS, Jakubiec WM, Kumar V, Silvia AM, Paige D, Dimitrova D, Li X, Ladutko L, Campbell S, Friedland G, Mitton-Fry M, Miller PF. Pharmacokinetics and whole-blood bactericidal activity against Mycobacterium tuberculosis of single doses of PNU-100480 in healthy volunteers. J Infect Dis. 2010 Sep 1;202(5):745-51. doi: 10.1086/655471. PMID 20629533
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1171001&StudyName=Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Study%20Of%20Single%20Doses%20Of%20PNU-100480%20In%20Healthy%20Adults